CLINICAL TRIAL: NCT03168425
Title: A Randomized Controlled Trial to Improve Discharge Opioid Prescribing After Cesarean Delivery
Brief Title: Opioid Prescribing After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Osmundson, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSMUNDSS04192017181235
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Surgery; Opioid Use
Keywords: safe opioid prescribing

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either a personalized prescribing algorithm based off of inpatient opioid use versus standard discharge opioid prescribing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored (Experimental): Participants will be prescribed an opioid based on a formula derived from inpatient opioid use
  Interventions: Other: Tailored prescription
- Control (Other): Participants will be prescribed 30 tablets of oxycodone 5mg, which is the average prescription currently given to our population.
  Interventions: Other: Control

INTERVENTIONS:
Other: Tailored prescription — Participants will be prescribed an opioid tablet number based on a formula derived from inpatient opioid use
  Arms: Tailored
Other: Control — Participants will be prescribed 30 tablets of oxycodone 5mg
  Arms: Control

SUMMARY:
The number of opioid overdose deaths in the United States has quadrupled in 15 years, a dramatic manifestation of the current opioid abuse epidemic. This rise parallels a sharp increase in the amount of legal prescription opioids dispensed. The abundance of prescription opioids available is a primary pathway for opioid abuse and diversion. Adjusting post- cesarean delivery opioid prescribing practices to better match actual patient need has the potential to reduce unused opioids available for diversion, nonmedical use, and development of chronic dependence, as well as reduce wasted resources.

DETAILED DESCRIPTION:
Preliminary data from a quality improvement project performed in our department found that most women are prescribed opioids after discharge that were significantly in excess of the actual opioids used. However there is a subset of women (~25%) who use all opioids and complain that they were not prescribed enough. The only variable predictive of post- discharge opioid use was Inpatient opioid use. These data were used to develop a formula for estimating outpatient use based on inpatient use. Currently there are no guidelines for outpatient prescribing either at our institution or on a national level. On average, most patients at our institution received 30 tablets of 5mg oxycodone at discharge. In surveying providers, very few looked at inpatient use and most had a standard prescription that they gave everyone.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-50 years old
* Women undergoing cesarean delivery at a single institution

Exclusion Criteria:

* Major post-surgical complications: cesarean hysterectomy, bowl or bladder injury, reoperation, ICU admission, wound infection or separation
* Chronic opioid use: Taking buprenorphine during pregnancy, taking an opioid for > 7 days during pregnancy.
* Non English or Spanish speaking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 190 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Osmundson, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osmundson SS, Raymond BL, Kook BT, Lam L, Thompson EB, Schornack LA, Voorhees CE, Richardson MG. Individualized Compared With Standard Postdischarge Oxycodone Prescribing After Cesarean Birth: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):624-630. doi: 10.1097/AOG.0000000000002782. PMID 30095773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tailored | Control
Started | 94 | 96
Completed | 87 | 85
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 5 | 8
Not completed — unable to confirm post op opioids | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored | Control | Total
Number analyzed (Participants) | 94 | 96 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 7 tailored/ 11 control subjects lost to follow-up
  years
    number analyzed (Participants) | 87 | 85 | 172
    (all) | 29.4 (5.9) | 30.4 (5.8) | 30.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 7 Tailored/ 11 control subjects lost to follow-up
  Participants
    number analyzed (Participants) | 87 | 85 | 172
    Female | 87 | 85 | 172
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 11 Tailored/ 7 control subjects were lost to follow-up
  Participants
    number analyzed (Participants) | 87 | 85 | 172
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 6 | 1 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 18 | 9 | 27
    White | 53 | 60 | 113
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 10 | 15 | 25
Region of Enrollment [Number; unit: participants] — Population: 7 Tailored/ 11 Control subjects lost to follow-up
  participants
    United States: number analyzed (Participants) | 87 | 85 | 172
    United States | 87 | 85 | 172

OUTCOME MEASURES:

1. Primary Outcome: Unused Opioids
Description: oxycodone 5mg tablet leftover from prescription at discharge
Time Frame: 4 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: oxycodone 5mg tablets
Groups:
- Tailored: Participants will be prescribed an opioid based on a formula derived from inpatient opioid use
  Participants who received an individualized prescription were discharged with 14 [interquartile range 12-16] oxycodone 5mg tablets.
Arm/Group | Tailored | Control
Number analyzed (Participants) | 87 | 85
oxycodone 5mg tablets | 5 [1 to 8] | 10 [0 to 22]

2. Secondary Outcome: Pain: Frequency That Participants Reported Uncontrolled Pain
Description: Frequency that participants reported uncontrolled pain
  Pain scores were examined based on how many negative responses indicating worse pain were reported to the five questions relating to analgesic adequacy. Thus participants could have a score that ranged from 0 to 5.
  Question 1 - I was discharged with too few opioid pills (Yes=1, No=0) Question 2 - Overall, my pain is poorly controlled by these medications (Yes=1, No=0) Question 3 - Overall, my pain from delivery has been worse than expected (Yes=1, No=0) Question 4 - Pain interfered significantly with my ability to do normal activities (Yes=1, No=0) Question 5 - Since discharge, I needed more opioid than what was expected (Yes=1, No=0)
Time Frame: 4 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tailored | Control
Number analyzed (Participants) | 87 | 85
score on a scale | 4 [2 to 5] | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Tailored | Control
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/96
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/96
Other Adverse Events (participants affected / at risk) | 0/94 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored (N=94) | Control (N=96)
Surgical Site Infection (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT03168425/Prot_SAP_000.pdf